CLINICAL TRIAL: NCT06802653
Title: Investigation on the Prevalence and Etiology of Adolescent Idiopathic Scoliosis in Nanchang Region
Status: Not yet recruiting | Type: Observational
Sponsor: Nanchang University Affiliated Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Wentao Zeng, YING Liang, Nanchang University Affiliated Rehabilitation Hospital
Other Study IDs: SFYLL-KY-PJ-2024-057
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-03

CONDITIONS: Scoliosis Idiopathic Adolescent
Keywords: scoliosis; screening; adolescents; prevalence; cost of screening
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: not provided

SUMMARY:
The purpose of this study is to investigate the prevalence and etiology of adolescent idiopathic scoliosis in the Nanchang region. Elementary and middle school students who met the inclusion criteria were included in the study and school-based scoliosis screening was conducted. Diagnosis of suspected scoliosis was determined by physical examination, Adams forward bend test, measurement of trunk rotation angle, and Standing Anteroposterior X-ray of the Spine. The prevalence of suspected scoliosis among elementary and middle school students was calculated. At the same time, the researchers kept detailed records of all costs incurred in the school screening.

DETAILED DESCRIPTION:
Scoliosis is a three-dimensional structural deformity of the spine that includes lateral curvature of the spine in the coronal plane, rotation in the horizontal plane, and alteration of the physiologic curvature in the sagittal plane. Scoliosis has an insidious onset and is often overlooked as there are no obvious symptoms in the early stages. As the disease progresses, it may lead to physical deformities, low back pain, decreased cardiorespiratory function, and may also cause psychological problems such as anxiety and depression. According to statistics, the global prevalence of scoliosis is 2-3%, and adolescent scoliosis is the most common type of scoliosis. The prevalence of scoliosis in adolescent females is higher than that of males. In recent years, the incidence of scoliosis has been on the rise as primary and secondary school students experience increased academic pressure and reduced physical activity and sleep time, which has caused great concern in society.

Scoliosis is thought to be associated with a variety of risk factors, including low BMI, gender differences, racial differences, asymmetrical backpack carrying, low physical activity, and prolonged screen viewing. However, despite the identification of many factors contributing to scoliosis, the comprehensive pathogenesis and natural progression of scoliosis are unknown.

Delaware pioneered school-based scoliosis screening in the 1960s, and it has since gradually spread throughout the United States, Canada, and Europe. Most studies have shown that early scoliosis screening is an effective way to prevent the progression of scoliosis in adolescents and reduce surgery rates. However, the implementation of mandatory scoliosis screening is controversial. Opponents of school-based scoliosis screening programs argue that, from a public health perspective, adolescent idiopathic scoliosis screening programs are not supported by sufficient evidence; from an economic perspective, school-based scoliosis screening requires a significant investment in human, material, and financial resources, and school-based scoliosis screening programs have not demonstrated significant cost-effectiveness.

The objectives of this study were to screen the prevalence of scoliosis among primary and secondary school students.

Study population Inclusion criteria: adolescents aged 9 to 14 years in primary and secondary schools.Exclusion criteria: congenital scoliosis, traumatic scoliosis, spinal tuberculosis, and other diseases caused by scoliosis.

Screening Methods In this study, 400 adolescents aged 9-12 years (from selected elementary schools) and 13-14 years (from middle schools) in Nanchang were screened. Prior to the assessment, basic information of the participants (including age, sex, height, weight, BMI, and medical history) was collected. Professional rehabilitation therapists evaluated the participants' posture and spinal rotation angles to determine the presence of scoliosis. Participants suspected of having scoliosis underwent further anteroposterior and lateral X-ray examinations for confirmation. Researchers collected data from the anteroposterior and lateral X-rays, including Cobb angle, Risser grade, Nash-Moe grade, and curve type. For participants diagnosed with scoliosis, additional parameters such as plantar pressure distribution, balance function, and respiratory function were collected.

① Plantar Pressure Measurement The specific procedure is as follows: The Footscan high-frequency plantar pressure distribution system (Belgium) was used. Participants stood barefoot on the pressure plate with their feet shoulder-width apart, looking at a target 1 meter ahead. Their arms hung naturally at their sides, and they breathed normally. After maintaining a stable posture for approximately 1 minute, the pressure sensor readings were recorded. Due to variations in height and body weight, the pressure data collected in this study were expressed as percentages of total plantar pressure. The selected parameters included total pressure on the left foot, total pressure on the right foot, forefoot pressure on both sides, and hindfoot pressure on both sides.

②Standard Posture Assessment

The specific procedure is as follows: The participant stood bareback with feet shoulder-width apart, eyes looking straight ahead, arms hanging naturally, and palms facing inward. The following were assessed:

1. Whether the shoulders were level;
2. Whether the scapulae were symmetrical;
3. Whether the inferior angles of the scapulae were at the same level;
4. Whether the lumbar concavities were symmetrical;
5. Whether the spinous process line was centered.

   * Adams Forward Bend Test The specific procedure is as follows: The participant stood upright with knees straight and feet together, then slowly bent forward to approximately 90° with arms extended and palms joined, gradually placing the hands between the knees. During this process, the examiner observed whether the participant's back showed any asymmetry or unevenness.

     * Angle of Trunk Rotation (ATR) Measurement A scoliometer was used to measure the degree of spinal rotation during the forward bend test. A reading greater than 5° was considered positive.

       * Standing Anteroposterior X-ray of the Spine The specific procedure is as follows: For patients of normal build, the X-ray settings were typically 120 kV, 200 mA, and 1 second. All patients underwent standing anteroposterior X-rays with feet shoulder-width apart, knees naturally extended, facing the X-ray tube, and hands raised with palms forward. If the leg length discrepancy exceeded 2 cm, the shorter side was elevated to keep the pelvis level. The central axis of the X-ray beam was aligned as closely as possible with the sagittal midline of the spine. A measurement scale was placed appropriately. A Cobb angle greater than 10° was diagnostic of scoliosis.

ELIGIBILITY:
Inclusion Criteria**

1. Age 9-14 years old, enrolled in elementary or middle school.
2. Local residents of Nanchang, excluding students from special schools for children with physical or intellectual disabilities.
3. No underlying medical conditions, and able to complete all examinations without difficulty.
4. Willing to participate in the screening and having signed an informed consent form.

Exclusion Criteria

1. Severe Medical Conditions: Individuals with severe diseases of the heart, liver, kidneys, endocrine system, or hematopoietic system.
2. Neurological or Psychiatric History: Individuals with a history of neurological or psychiatric disorders.
3. Refusal to Participate: Individuals who are unwilling or refuse to participate in the screening.
4. Severe Osteoporosis: Individuals diagnosed with severe osteoporosis.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: adolescents aged 9 to 14 years in primary and secondary schools
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Footscan Plantar Pressure Test Parameters | The process from enrollment to the completion of screening takes about one week.
  The results of the Footscan plantar pressure test parameters for participants included total pressure on the left foot, total pressure on the right foot, forefoot pressure on both sides, and hindfoot pressure on both sides.
Physical Examination | The process from enrollment to the completion of screening takes about one week.
  The examinee has a bare back, stands naturally, feet shoulder-width apart, eyes flat, arms down, palms facing inward. The examiner observes whether the patient's shoulders are equal in height; whether the angles of both subscapularis are at the same level; whether the lumbar concavity is symmetrical on both sides; whether the iliac crests are equal in height bilaterally; and whether the spinous processes are deviating from the median axis.
standing anteroposterior X-rays of the spine | The process from enrollment to the completion of screening takes about one week.
  Information from standing anteroposterior X-rays of the spine, including Cobb angle, Risser grade, Nash-Moe grade, and curve type
participants' basic information | The process from enrollment to the completion of screening takes about one week.
  basic information from participants, including age, sex, height, weight, BMI, and medical history.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchang University Affiliated Rehabilitation Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Yes